CLINICAL TRIAL: NCT06993376
Title: Comparison Between the Ultrasound Guided Pericapsular Nerve Group Block and Erector Spinae Plane Block on Motor Power Postoperative in Elderly Patients Undergoing Total Hip Replacement Surgeries; A Randomized Controlled Trial
Brief Title: PENG Block vs ESPB in Elderly Undergoing Hip Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdelghany ali, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N22-2023/MD
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia for Hip Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Active Comparator)
  Interventions: Procedure: PENG block
- ESPb (Active Comparator)
  Interventions: Procedure: ESPB

INTERVENTIONS:
Procedure: PENG block — Group LESBP: 28 patients will receive single shot LESPB after spinal induction. Group PENG: 28 patients will receive single shot PENG after spinal induction.
  Arms: PENG block
Procedure: ESPB — Group LESBP: 28 patients will receive single shot LESPB after spinal induction. Group PENG: 28 patients will receive single shot PENG after spinal induction.
  Arms: ESPb

SUMMARY:
To our knowledge, the comparison between the ultrasound-guided lumbar erector spinae plane block and the pericapsular nerve group block has not been investigated before in previous literature.

ELIGIBILITY:
Inclusion Criteria:

* Both genders Type of surgery; unilateral elective total hip replacement. Physical status ASA I, II Age more than or equal 65 Years. Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Patient refusal. Patients with known sensitivity or contraindication to drugs used in the study (local anesthetics & opioids).

History of psychological disorders and/or chronic pain. Pre- existing peripheral neuropathies Coagulopathy. Infection of the skin at the site of needle puncture area.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor power | 24 hours postoperative
  The result of substraction of VAS from MRC at ipsilateral lower limb at the time of regaining of full motor power in the contralateral lower limb (delta).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol